CLINICAL TRIAL: NCT01533688
Title: Efficacy and Tolerability of Various Bowel Preparations in Diabetic Patients: A Randomized Controlled Trial
Brief Title: Study of Efficacy and Tolerability of Various Bowel Preps in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2869
Record Dates: First submitted 2012-01-19; First posted 2012-02-15 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Golytely; Bisacodyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Golytely + placebo (Active Comparator): 4 liters of polyethylene glycol electrolyte lavage solution (PEG-ELS-(GoLytely)+ placebo pill
  Interventions: Drug: Golytely (polyethylene glycol electrolyte lavage solution) and placebo
- Golytely Split + placebo (Placebo Comparator): split dose(2 L day before procedure and 2 L day of procedure) of 4 liters of Golytely + placebo pill
  Interventions: Drug: split dose of Golytely (polyethylene glycol electrolyte lavage solution) + placebo
- Golytely Split + Bisacodyl (Experimental): split dose (2 L day prior to procedure and 2 L day of procedure) of 4 liters of Golytely + bisacodyl 10 mg
  Interventions: Drug: split dose of Golytely (polyethylene glycol electrolyte lavage solution) and bisacodyl

INTERVENTIONS:
Drug: Golytely (polyethylene glycol electrolyte lavage solution) and placebo — 4 liters of polyethylene glycol electrolyte lavage solution (PEG-ELS-(GoLytely))+ placebo given the evening prior to the colonoscopy
  Arms: Golytely + placebo
Drug: split dose of Golytely (polyethylene glycol electrolyte lavage solution) + placebo — split dose (2 L taken the evening before and 2 L taken the morning of the colonoscopy) of 4 liters Golytely + placebo
  Arms: Golytely Split + placebo
Drug: split dose of Golytely (polyethylene glycol electrolyte lavage solution) and bisacodyl — split dose ( 2 L taken the evening before and 2 L taken the morning of the colonoscopy) of 4 liters of Golytely + bisacodyl 10 mg
  Arms: Golytely Split + Bisacodyl

SUMMARY:
Poor bowel preparation and patient intolerance of the procedure are the most important factors contributing to the limitation of colonoscopy. Inadequate bowel cleansing results in incomplete testing, increased potential to miss lesions, increased cost, and decreased patient satisfaction. The investigators hope to gain better insight into which bowel preparation works best in diabetic patients and hence would increase patient satisfaction, tolerability of the bowel preparation and decrease overall costs. The investigators will investigate which bowel preparation for colonoscopy will work optimally in diabetic patients using three different regimens.

ELIGIBILITY:
Inclusion Criteria:

* adult diabetic outpatients referred for elective colonoscopy

Exclusion Criteria:

* patients < 18 years of age or > 75 yrs of age,
* known or suspected pregnancy,
* known or suspected renal failure,
* unstable angina,
* acute coronary syndrome,
* decompensated congestive heart failure,
* decompensated liver failure,
* known or suspected bowel obstruction,
* major psychiatric illness,
* solid organ transplant patients,
* known allergies to PEG-ELS or bisacodyl,
* prior alimentary tract surgery or refusal to consent to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Madhoun, MD, Principal Investigator — University of Oklahoma Health Science Center
Locations (1):
- Oklahoma VA Medical Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Golytely + Placebo | Golytely Split + Placebo | Golytely Split + Bisacodyl
Started | 71 | 70 | 71
Completed | 63 | 60 | 63
Not Completed | 8 | 10 | 8
Not completed — Withdrawal by Subject | 5 | 4 | 3
Not completed — Medically unstable | 1 | 3 | 3
Not completed — Had colonoscopy at outside hospital | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golytely + Placebo | Golytely Split + Placebo | Golytely Split + Bisacodyl | Total
Number analyzed (Participants) | 63 | 60 | 63 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.4) | 62.8 (7.2) | 63.2 (6.7) | 63.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 61 | 59 | 58 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White race | 41 | 45 | 51 | 137
  Other | 22 | 15 | 12 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 60 | 63 | 186

OUTCOME MEASURES:

1. Primary Outcome: Measure the % of Participants With Effective (How Well the Colon is Cleansed Using the Validated Boston Bowel Preparation Scale) for Various Bowel Preparations for Colonoscopy.
Description: The investigators will measure the number/% of participants who will have good to excellent bowel preparations defined by the Boston Bowel Prep Scale(BBPS) with a score of 6 or more, rated by blinded colonoscopist.
Time Frame: Day 1
Population: We have missing data regarding reporting of Boston bowel preparation scores (BBPS), some providers didn't provide the BBPS and provided only subjective assessment of the bowel preparation (for example, good or excellent)
Measure: Count of Participants; unit: Participants
Arm/Group | Golytely + Placebo | Golytely Split + Placebo | Golytely Split + Bisacodyl
Number analyzed (Participants) | 63 | 60 | 63
Participants | 42 | 50 | 47

2. Secondary Outcome: Measure of Patients Who Develop (Tolerance)Side Effects of Taking Bowel Preparations.
Description: Number of Participants Who Developed Side Effects of Taking Bowel Preparations
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Groups:
- Golytely Split+Placebo: split dose(2 L day before procedure and 2 L day of procedure) of 4 liters of Golytely + placebo pill
  split dose of Golytely (polyethylene glycol electrolyte lavage solution) + placebo: split dose (2 L taken the evening before and 2 L taken the morning of the colonoscopy) of 4 liters Golytely + placebo
- Golytely Split+Bisacodyl: split dose (2 L day prior to procedure and 2 L day of procedure) of 4 liters of Golytely + bisacodyl 10 mg
  split dose of Golytely (polyethylene glycol electrolyte lavage solution) and bisacodyl: split dose ( 2 L taken the evening before and 2 L taken the morning of the colonoscopy) of 4 liters of Golytely + bisacodyl 10 mg
Arm/Group | Golytely + Placebo | Golytely Split+Placebo | Golytely Split+Bisacodyl
Number analyzed (Participants) | 63 | 60 | 63
Participants | 24 | 28 | 28

ADVERSE EVENTS:
Arm/Group | Golytely + Placebo | Golytely Split + Placebo | Golytely Split + Bisacodyl
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 24/63 | 27/60 | 28/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golytely + Placebo (N=63) | Golytely Split + Placebo (N=60) | Golytely Split + Bisacodyl (N=63)
nausea and vomiting (Gastrointestinal disorders) | 6 | 4 | 6
Bloating (Gastrointestinal disorders) | 10 | 10 | 10
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 2
Rectal burning sensation (Gastrointestinal disorders) | 6 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No